CLINICAL TRIAL: NCT06117579
Title: Effect of Inspiratory Muscle Training on Daytime Sleepiness in Obstructive Sleep Apnea Syndrome : Prospective Randomized Controlled Trial
Brief Title: Effect of Inspiratory Muscle Training in Obstructive Sleep Apnea Syndrome.
Acronym: NOCTURNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2023-08
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive Sleep Apnea; Inspiratory muscle training
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (Experimental): Step 1:
  During the consultation to diagnose obstructive sleep disorder with the pulmonologist (following polysomnography) to set up continuous positive airway pressure (CPAP):
  * Introduction of CPAP
  * Epworth Sleepiness Scale (ESS)
  * Maximum Inspiratory Pressure (MIP) measurement
  * Explanation of exercise program and use of POWERBreathe
  Step 2:
  6-week telephone follow-up with measurement of Epworth Sleepiness Scale (ESS)
  Step 3:
  Follow-up visit at 12 weeks after introduction of CPAP:
  * Review of CPAP implementation
  * Epworth Sleepiness Scale (ESS)
  * MIP measurement
  Interventions: Other: Inspiratory muscle training
- Control group (No Intervention): Step 1:
  During the consultation to diagnose obstructive sleep disorder with the pulmonologist (following polysomnography) to set up continuous positive airway pressure (CPAP):
  * Introduction of CPAP
  * Epworth Sleepiness Scale (ESS)
  * Maximum Inspiratory Pressure (MIP) measurement
  Step 2:
  6-week telephone follow-up with measurement of Epworth Sleepiness Scale (ESS)
  Step 3:
  Follow-up visit at 12 weeks after introduction of CPAP:
  * Review of CPAP implementation
  * Epworth Sleepiness Scale (ESS)
  * MIP measurement

INTERVENTIONS:
Other: Inspiratory muscle training — Description of a typical session:
  Session duration: between 12 and 20 minutes 3 cycles of 30 repetitions with 1 minute of break between each cycle. The patient should inhale as hard as possible against an inspiratory resistance generated by a valve device.
  Arms: Inspiratory muscle training group

SUMMARY:
Sleep apnea-hypopnea syndrome is a sleep-related respiratory disorder characterized by partial or total interruptions in breathing during sleep. The majority of syndromes involve an obstructive mechanism (OSA), caused by a reduction in the caliber of the upper airway (UA), most often associated with hypotonia of the surrounding muscles, preventing air from entering the UA during inspiration. The clinical consequences of this syndrome are excessive fatigue and daytime sleepiness, which have a negative impact on the quality of life of patients.

Despite the positive results on apnea-hypopnea index and daytime sleepiness of continuous positive airway pressure (today's reference treatment), its 3-year compliance rate (i.e 59.9% according to a study by Abdelghani et al points to the need to develop other associated therapies.

Several studies have demonstrated the efficacy of physiotherapy, such as physical activity and oro-pharyngeal muscle strengthening, notably on the apnea-hypopnea index and daytime sleepiness measured by the Epworth scale.

Few studies have investigated the effect of inspiratory muscle training (IMT), even though the use of the inspiratory musculature (i.e. the diaphragm) is a means of supplementing the peri-pharyngeal muscles, as it helps to maintain the permeability of the upper airways. Inspiratory muscle training (IMT) could therefore be considered as part of the physiotherapeutic management of the OSA. The heterogeneity of current results concerning IMT in OSA , but above all the lack of evidence that it is dangerous, means that new clinical studies could be carried out in an attempt to demonstrate its efficacy. Our research hypothesis is therefore as follows: Implementing an inspiratory muscle strengthening protocol in patients suffering from OSA can reduce daytime sleepiness.

DETAILED DESCRIPTION:
Sleep apnea-hypopnea syndrome is a sleep-related respiratory disorder characterized by partial or total interruptions in breathing during sleep. The majority of syndromes involve an obstructive mechanism (OSA), caused by a reduction in the caliber of the upper airway (UA), most often associated with hypotonia of the surrounding muscles, preventing air from entering the UA during inspiration. The clinical consequences of this syndrome are excessive fatigue and daytime sleepiness, which have a negative impact on the quality of life of patients.

Despite the positive results on apnea-hypopnea index and daytime sleepiness of continuous positive airway pressure (today's reference treatment), its 3-year compliance rate (i.e 59.9% according to a study by Abdelghani et al points to the need to develop other associated therapies.

Several studies have demonstrated the efficacy of physiotherapy, such as physical activity and oro-pharyngeal muscle strengthening, notably on the apnea-hypopnea index and daytime sleepiness measured by the Epworth scale.

Few studies have investigated the effect of inspiratory muscle training (IMT), even though the use of the inspiratory musculature (i.e. the diaphragm) is a means of supplementing the peri-pharyngeal muscles, as it helps to maintain the permeability of the upper airways. Inspiratory muscle training (IMT) could therefore be considered as part of the physiotherapeutic management of the OSA. The heterogeneity of current results concerning IMT in OSA , but above all the lack of evidence that it is dangerous, means that new clinical studies could be carried out in an attempt to demonstrate its efficacy. Our research hypothesis is therefore as follows: Implementing an inspiratory muscle strengthening protocol in patients suffering from OSA can reduce daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age with
* OSA with an Apnea Hypopnea Index ≥ 5 requiring CPAP

Exclusion Criteria:

* Sleep apnea of neurological or mixed origin,
* Contraindication to or refusal of CPAP,
* Cognitive disorders,
* protected persons (under guardianship or curatorship),
* persons under court protection,
* persons not affiliated to a social security scheme
* pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Change in Daytime sleepiness | 12 weeks
  Change in daytime sleepiness measured by the Epworth Sleepiness Scale following the introduction of IMT combined with CPAP Epworth Sleepiness Scale ranged from 0 (it is unlikely that you are abnormally sleepy) to 24 (you are excessively sleepy and should consider seeking medical attention).

CONTACTS AND LOCATIONS:
Overall Officials: Marie DEVAUX, Dr, Principal Investigator — CHU d'Orléans
Locations (1):
- Chu Orleans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou KT, Tsai YL, Yeh WY, Chen YM, Huang N, Cheng HM. Risk of work-related injury in workers with obstructive sleep apnea: A systematic review and meta-analysis. J Sleep Res. 2022 Feb;31(1):e13446. doi: 10.1111/jsr.13446. Epub 2021 Aug 12. PMID 34384138
- [Background] Sabil A, Bignard R, Gerves-Pinquie C, Philip P, Le Vaillant M, Trzepizur W, Meslier N, Gagnadoux F. Risk Factors for Sleepiness at the Wheel and Sleep-Related Car Accidents Among Patients with Obstructive Sleep Apnea: Data from the French Pays de la Loire Sleep Cohort. Nat Sci Sleep. 2021 Oct 5;13:1737-1746. doi: 10.2147/NSS.S328774. eCollection 2021. PMID 34675722
- [Background] Peng J, Yuan Y, Zhao Y, Ren H. Effects of Exercise on Patients with Obstructive Sleep Apnea: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2022 Aug 31;19(17):10845. doi: 10.3390/ijerph191710845. PMID 36078558
- [Background] Abdelghani A, Slama S, Hayouni A, Harrabi I, Mezghanni S, Garrouche A, Klabi N, Benzarti M, Jerray M. [Acceptance and long-term compliance to continuous positive airway pressure in obstructive sleep apnea. A prospective study on 72 patients treated between 2004 and 2007]. Rev Pneumol Clin. 2009 Jun;65(3):147-52. doi: 10.1016/j.pneumo.2009.03.010. Epub 2009 Jun 3. French. PMID 19524803
- [Background] Azeredo LM, Souza LC, Guimaraes BLS, Puga FP, Behrens NSCS, Lugon JR. Inspiratory muscle training as adjuvant therapy in obstructive sleep apnea: a randomized controlled trial. Braz J Med Biol Res. 2022 Oct 3;55:e12331. doi: 10.1590/1414-431X2022e12331. eCollection 2022. PMID 36197415
- [Background] Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med. 2013 Oct 15;188(8):996-1004. doi: 10.1164/rccm.201303-0448OC. PMID 23721582